CLINICAL TRIAL: NCT03435913
Title: Assessment of Transpulmonary Driving Pressure and Intra-abdominal Pressure Relationship at Different Levels of Positive End-expiratory Pressure (PEEP) During Laparoscopic Surgery
Brief Title: Transpulmonary Driving Pressure and Intra-abdominal Pressure Relationship During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Anesthesiology Consultant, Hospital Universitario La Fe
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/0602
Record Dates: First submitted 2018-01-30; First posted 2018-02-19 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia, General/Methods; Laparoscopy; Respiration, Artificial; Positive-Pressure Respiration; End-Expiratory Pressure, Positive; Ventilator-Induced Lung Injury
Keywords: Mechanical ventilation; Driving Pressure; Protective Lung VEntilation
MeSH Terms: conditions — Respiratory Aspiration; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PEEP ventilation (Experimental): During pneumoeperitoneum insufflation the patient is ventilated with 7 ml/kg per ideal body weight, inspiration:expiration (I:E) ratio 1:2, and respiration rate (RR) to maintain EtCO2 at 35-38 mmHg and 5 cmH20 of PEEP at every intra-abdominal pressure (IAP) step (8, 12 and 15 mmHg).
  Interventions: Other: Standard PEEP ventilation; Other: Matched PEEP ventilation
- Matched PEEP Ventilation (Experimental): During pneumoeperitoneum insufflation the patient is ventilated with 7 ml/kg per ideal body weight, inspiration:expiration (I:E) ratio 1:2, and respiration rate (RR) to maintain EtCO2 at 35-38 mmHg and a level of PEEP matched to every IAP step (8, 12 and 15 mmHg).
  1 mmHg = 1,36 cmH20.
  Between the standard and matched PEEP intervention there is a washout period that with a recruitment maneuver to re-establish baseline lung condition.
  Interventions: Other: Standard PEEP ventilation; Other: Matched PEEP ventilation

INTERVENTIONS:
Other: Standard PEEP ventilation — During mechanical ventilation a fixed PEEP (5 mcH2O) is set at all IAP levels during pneumoperitoneum insufflation
Other: Matched PEEP ventilation — During mechanical ventilation PEEP is matched to IAP level

SUMMARY:
Objective: The aim of this project is to evaluate how intra-abdominal pressure paired coupled with different ventilatory positive end-expiratory pressure levels affects the transpulmonary driving pressure during pneumoperiteneum insufflation for laparoscopic surgery.

Methodology: Patients undergoing laparoscopic surgery will be included. The study will investigate the relationship between intra-abdominal pressure (IAP) and transpulmonary driving pressure (TpDp) and the effect of titration of PEEP on their relationship.

At three different levels of intra-abdominal pressure, the respiratory driving pressure (RDp) and TpDp in each subject will be measured in each subject. The same subject will undergo two different ventilation strategies. Demographic data (height, weight, body mass index and sex), ASA physical status (surgical risk classification of the American Society of Anesthesiology), number of previous abdominal surgeries, number of previous pregnancies, and respiratory comorbidities will be collected. Respiratory pressures and mechanics will be recorded at each level of intra-abdominal pressure (IAP) during each ventilatory strategy. The variables recorded will include: airway pressures (Plateau pressure Pplat, Peak pressure, Ppeak), the final esophageal pressure of inspiration and expiration and pulmonary stress index. Mixed linear regression will be used to evaluate the relationship between different PEEP levels, IAP and TpDp by adjusting for known confounders and adding individuals as a random factor. Likewise, an analysis using a mixed linear regression model with the pulmonary stress index as a function of the intra-abdominal pressure, the ventilation regime, and a specific random intercept term for each subject will be performed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) risk scale I to III
* Age > 18 years
* Previously signed informed consent
* Undergoing laparoscopic surgery

Exclusion Criteria:

* ASA ≥ IV
* Pregnancy
* Advanced liver, kidney or cardiopulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Transpulmonary driving pressure (TpDp) difference between standard and matched PEEP ventilation | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  TpDp (assessed in centimeters of water, cmH20) as assessed by ventilatory pressure and pleural pressure (recorded by an esophageal probe) is recorded at every intra-abdominal pressure level during pneumoperitoneum insufflation. The primary outcome is the difference between a standard perioperative management (fixed PEEP + 15 mmHg pneumoperitoneum pressure) and matched PEEP to intra-abdominal pressure and 8mmHg intra-abdominal pressure

SECONDARY OUTCOMES:
Transpulmonary driving pressure and intra-abdmominal pressure relationship (multivariate adaptive linear regression) | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  TpDp (in cmH20) is recorded at different levels of IAP and with two different PEEP settings (in cmH20; two levels are: fixed at each IAP level, standard group and matched at each IAP level, matched group). The relationship between TpDp and IAP (both treated as continuous variables) at each PEEP level is plotted and a multiadaptive linear regression is fitted.
Transpulmonary driving pressure and respiratory driving pressure (RDp) relationship (multivariate adaptive linear regression). | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  Respiratory driving pressure (transpulmonary driving pressure + pressure to move the chest wall, in cmH20, RpDp) and TpDp relationship at each IAP and PEEP level will be assessed. The relationship between TpDp and RpDp (both treated as continuous variables) at each PEEP level is plotted and a multiadaptive linear regression is fitted.
Respiratory system compliance (Crs) difference between standard and matched PEEP levels | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  Respiratory system compliance measures the system's ability to stretch. It has two components Lung and Chest Wall (measured in milliliter/centimeters of water, ml/cmH20)
Pulmonary compliance (Cp) difference | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  Respiratory system compliance measures the system's ability to stretch (ml/cmH20). It has two components Lung and Chest Wall (measured in milliliter/centimeters of water, ml/cmH20). By using an esophageal probe measurement the two can be partitioned and analyzed separately.
Chest wall compliance (CCw) difference | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  Respiratory system compliance measures the system's ability to stretch (ml/cmH20). It has two components Lung and Chest Wall (measured in milliliter/centimeters of water, ml/cmH20). By using an esophageal probe measurement the two can be partitioned and analyzed separately.
Pulmonary Stress index difference | Pneumoperitoneum insufflation before surgery (up to 30 minutes)
  Stress index is based on respiratory pressure curve analysis and assess whether the lungs are overdistended or collapsed

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Background] Cortes-Puentes GA, Gard KE, Adams AB, Faltesek KA, Anderson CP, Dries DJ, Marini JJ. Value and limitations of transpulmonary pressure calculations during intra-abdominal hypertension. Crit Care Med. 2013 Aug;41(8):1870-7. doi: 10.1097/CCM.0b013e31828a3bea. PMID 23863222
- [Background] Cinnella G, Grasso S, Spadaro S, Rauseo M, Mirabella L, Salatto P, De Capraris A, Nappi L, Greco P, Dambrosio M. Effects of recruitment maneuver and positive end-expiratory pressure on respiratory mechanics and transpulmonary pressure during laparoscopic surgery. Anesthesiology. 2013 Jan;118(1):114-22. doi: 10.1097/ALN.0b013e3182746a10. PMID 23196259
- [Background] D'Antini D, Rauseo M, Grasso S, Mirabella L, Camporota L, Cotoia A, Spadaro S, Fersini A, Petta R, Menga R, Sciusco A, Dambrosio M, Cinnella G. Physiological effects of the open lung approach during laparoscopic cholecystectomy: focus on driving pressure. Minerva Anestesiol. 2018 Feb;84(2):159-167. doi: 10.23736/S0375-9393.17.12042-0. Epub 2017 Jul 5. PMID 28679201